CLINICAL TRIAL: NCT06863155
Title: Ultrathin Strut Sirolimus-eluting Stent With Bioabsorbable Polymer in Patients Receiving Chronic Oral Anticoagulation
Acronym: ACO_FLEX
Status: Recruiting | Type: Observational
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Other Study IDs: rEPIC13-ACO-FLEX
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Disease; Ischemic Heart Disease
Keywords: Chronic oral anticoagulation; Ultrathin-strut stent; Biodegradable polymer; High-bleeding risk; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Supraflex Cruz Sirolimus-eluting Stent
  Interventions: Device: Supraflex Cruz Sirolimus-eluting Stent

INTERVENTIONS:
Device: Supraflex Cruz Sirolimus-eluting Stent — PCI with SupraFlex Cruz® stent in de novo coronary stenosis of patients under chronic oral anticoagulation.

SUMMARY:
Patients receiving chronic oral anticoagulation with indication for percutaneous coronary revascularization with stent implantation, and needing for antiplatelet therapy, are at high risk of bleeding. The new generation of ultrathin strut sirolimus-eluting stent with bioabsorbable polymer allow for shorter antiplatelets regimens and could be a good option for this high-bleeding risk patients.

DETAILED DESCRIPTION:
Patients receiving chronic oral anticoagulation with indication for percutaneous coronary revascularization with stent implantation, and needing for antiplatelet therapy, are at high risk of bleeding. The new generation of ultrathin strut sirolimus-eluting stent with bioabsorbable polymer allow for shorter antiplatelets regimens and could be a good option for this high-bleeding risk patients.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all inclusion criteria:

* Patients with Signed informed consent and
* Patients with >=18 years old and
* Patients with chronically receiving oral anticoagulation treatment with any type of anticoagulant for any reason and
* Patients with de novo Coronary artery disease requiring both elective or urgent percutaneous revascularization due to stable coronary artery disease or acute coronary syndrome with or without ST-segment elevation, and in which an ultrathin strut Sirolimus-eluting stent with bioabsorbable polymer has been used

Exclusion Criteria:

Patients do not have to meet any exclusion criteria

* Patients treated percutaneously with any type of stent other than the SupraFlex Cruz® in the 6 months prior to the index procedure in which he or she is included.
* Use in the same procedure or in a scheduled procedure of other stents different from the one evaluated for the treatment of another vessel(s).
* Patients treatment for restenosis or stent thrombosis.
* Patients presentation in cardiogenic shock or after cardiorespiratory arrest.
* Patients with allergy to any of the components of the stent to be used.
* Patients with impossibility for follow-up.
* Patients with life expectancy less than 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients under chronic oral anticoagulation undergoing PCI with implantation of a SupraFlex Cruz(r) stent
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
NACE (Net Adverse Clinical Events) | 12 month
  Combined endpoint of Cardiac Death, Acute Myocardial Infarction, Stroke, Need for new Treated Vessel Revascularization (TVR) and BARC (Bleeding Academic Research Consortium) 3-5

SECONDARY OUTCOMES:
MACE (Major Adverse Cardiac Events) | 12 months
  To assess the occurrence of major adverse cardiac events (MACE) in patients receiving chronic oral anticoagulation who have been treated with ultrathin strut Sirolimus-eluting stents with bioabsorbable polymer.
MACE (Major Adverse Cardiac Events) | 6 months
  To assess the occurrence of major adverse cardiac events (MACE) in patients receiving chronic oral anticoagulation who have been treated with ultrathin strut Sirolimus-eluting stents with bioabsorbable polymer.
TLF (Target Lesion Failure) | 12 months
  To assess the failure rate of the lesion treated (TLF) with ultrathin strut Sirolimus-eluting stent with bioabsorbable polymer in patients receiving chronic oral anticoagulation.
TLF (Target Lesion Failure) | 6 months
  To assess the failure rate of the lesion treated (TLF) with ultrathin strut Sirolimus-eluting stent with bioabsorbable polymer in patients receiving chronic oral anticoagulation.
Death | 12 months
  To assess the occurrence of Death
Death | 6 months
  To assess the occurrence of Death
Acute Myocardial Infarction (AMI) | 12 months
  To assess the occurrence of AMI
Acute Myocardial Infarction (AMI) | 6 months
  To assess the occurrence of AMI
Stroke | 12 months
  To assess the occurrence of Stroke
Stroke | 6 months
  To assess the occurrence of Stroke
Target vessel revascularization (TVR) | 12 months
  To assess the occurrence of TVR
Target vessel revascularization (TVR) | 6 months
  To assess the occurrence of TVR

CONTACTS AND LOCATIONS:
Locations (8):
- Spain (8):
  - Hospital General Universitario de Albacete, Albacete
  - Hospital Universitario San Juan de Alicante, Alicante
  - Hospital General Universitario de Merida, Badajoz
  - Hospital General Universitari de Castelló, Castelló
  - H.G.U. de Ciudad Real., Ciudad Real
  - Hospital General Universitari d'Elx, Elche
  - Hospital Universitario Puerta de Hierro, Majadahonda
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza

REFERENCES:
- [Background] Lemos PA, Chandwani P, Saxena S, Ramachandran PK, Abhyankar A, Campos CM, Marchini JF, Galon MZ, Verma P, Sandhu MS, Parikh N, Bhupali A, Jain S, Prajapati J. Clinical outcomes in 995 unselected real-world patients treated with an ultrathin biodegradable polymer-coated sirolimus-eluting stent: 12-month results from the FLEX Registry. BMJ Open. 2016 Feb 17;6(2):e010028. doi: 10.1136/bmjopen-2015-010028. PMID 26888727
- [Background] Choudhury A, Garg S, Smith J, Sharp A, Nabais de Araujo S, Chauhan A, Patel N, Wrigley B, Chattopadhyay S, Zaman AG. Prospective evaluation of an ultrathin strut biodegradable polymer-coated sirolimus-eluting stent: 12 months' results from the S-FLEX UK registry. BMJ Open. 2019 Oct 11;9(10):e026578. doi: 10.1136/bmjopen-2018-026578. PMID 31604782
- [Background] Zaman A, de Winter RJ, Kogame N, Chang CC, Modolo R, Spitzer E, Tonino P, Hofma S, Zurakowski A, Smits PC, Prokopczuk J, Moreno R, Choudhury A, Petrov I, Cequier A, Kukreja N, Hoye A, Iniguez A, Ungi I, Serra A, Gil RJ, Walsh S, Tonev G, Mathur A, Merkely B, Colombo A, Ijsselmuiden S, Soliman O, Kaul U, Onuma Y, Serruys PW; TALENT trial investigators. Safety and efficacy of a sirolimus-eluting coronary stent with ultra-thin strut for treatment of atherosclerotic lesions (TALENT): a prospective multicentre randomised controlled trial. Lancet. 2019 Mar 9;393(10175):987-997. doi: 10.1016/S0140-6736(18)32467-X. Epub 2019 Feb 28. PMID 30827782
- [Background] Biscaglia S, Guiducci V, Escaned J, Moreno R, Lanzilotti V, Santarelli A, Cerrato E, Sacchetta G, Jurado-Roman A, Menozzi A, Amat Santos I, Diez Gil JL, Ruozzi M, Barbierato M, Fileti L, Picchi A, Lodolini V, Biondi-Zoccai G, Maietti E, Pavasini R, Cimaglia P, Tumscitz C, Erriquez A, Penzo C, Colaiori I, Pignatelli G, Casella G, Iannopollo G, Menozzi M, Varbella F, Caretta G, Dudek D, Barbato E, Tebaldi M, Campo G; FIRE Trial Investigators. Complete or Culprit-Only PCI in Older Patients with Myocardial Infarction. N Engl J Med. 2023 Sep 7;389(10):889-898. doi: 10.1056/NEJMoa2300468. Epub 2023 Aug 26. PMID 37634150
- [Background] Paradies V, Maurina M, Tonino P, Hofma SH, Vos J, van Kuijk JP, Oemrawsingh RM, Mafragi AA, Spano F, Pisters R, Polad J, Ijsselmuiden S, Cambero MM, Smits PC. Comparison of Supraflex Cruz 60 mum Versus Ultimaster Tansei 80 mum Stent Struts in High Bleeding Risk PCI Patients: Study design and Rational of Compare 60/80 HBR trial. Am J Cardiol. 2023 Nov 1;206:230-237. doi: 10.1016/j.amjcard.2023.08.046. Epub 2023 Sep 13. PMID 37708755